CLINICAL TRIAL: NCT05750511
Title: Prospective Multicenter Translational Study to Validate Molecular Biomarkers (TMB, PD-L1) on Pre-treatment Tumor Tissue as Predictors of Therapy Outcome in Metastatic Melanoma Patients
Brief Title: Multicenter Tissue Registry in Melanoma
Acronym: TRIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dermatologic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: CA209-578
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Metastatic Melanoma
Keywords: melanoma; biomarker; tumor tissue; systemic therapy; immune checkpoint therapy; targeted therapy; PD-L1; Tumor mutational burden
MeSH Terms: conditions — Melanoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — pre-treatment tumor tissue of different origin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metastatic melanoma: 1,000 subjects with metastatic melanoma stage III or IV suitable for systemic treatment from centers of the German Dermatologic Cooperative Oncology Group (DeCOG)
  Interventions: Diagnostic Test: molecular tissue analysis

INTERVENTIONS:
Diagnostic Test: molecular tissue analysis

SUMMARY:
The prospective multicenter translational study Tissue Registry in Melanoma (ADOREG/TRIM; CA209-578) aimed to validate the Tumor Mutational Burden (TMB) and the PD-L1 expression (PD-L1) from a pre-therapeutically obtained tumor tissue sample as a predictor of a subsequent systemic therapy in a large real-world cohort of metastatic melanoma patients.

DETAILED DESCRIPTION:
The aim of the present study is to identify and validate molecular and clinical biomarkers of therapy outcome in metastatic melanoma. Clinical and molecular parameters of melanoma patients and their tumors will be collected in an online-based registry (ADOREG), and thereafter correlated with the outcome of subsequent systemic therapies in terms of progression-free survival, overall survival, and treatment response. Systemic therapies will include all types of currently used regimens (kinase inhibitors, immune checkpoint inhibitors, chemotherapy). FFPE tissue samples will comprise different time points (primary tumors versus metastases) as well as tumor sites (lymph node versus organ metastases) to identify potential differences in the predictive value of these materials. The anticipated results from these analyses are of essential importance for future patient selection for individualized therapy strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed melanoma stage III or IV.
2. Clinically eligible for systemic cancer therapy (immune checkpoint inhibitors, targeted agents).
3. Tumor tissue biopsy already existing (metastasis tissue as recent as possible, but older tissue material or primary tumor tissue also possible).
4. Patient has given written informed consent for the current study as well as for his data to be entered into the ADOREG online database system.
5. Patient is ≥18 years old.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with metastatic melanoma stage III or IV suitable for systemic treatment
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
BOR | through study completion, an average of 1 year
  best overall response (BOR)
PFS | through study completion, an average of 1 year
  progression-free survival (PFS)
OS | through study completion, an average of 1 year
  overall survival (OS)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, MD, Study Chair — Dermatologic Cooperative Oncology Group
Locations (14):
- Germany (14):
  - Dept. of Dermatology, University Hospital Tuebingen, Tübingen, Baden-Wurttemberg
  - Department of Dermatology, ElbeKliniken - Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Department of Dermatology, The Saarland University Hospital, Homburg/Saar, Saarland
  - Dept. of Dermatology, University of Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Dept. of Dermatology, Helios Clinic Erfurt, Erfurt, Thuringia
  - Department of Dermatology, University Hospital, Augsburg
  - Department of Dermatology, University Hospital, Dresden
  - Department of dermatology, University Hospital, Essen
  - Medizinische Hochschule,dermatologische Klinik und Poliklinik, Hanover
  - Department of Dermatology, Ludwigshafen
  - Skin Cancer Unit, University Hospital, Mannheim
  - Department of Dermatology, University Hospital, Minden
  - Department of Dermatology, Oberhausen
  - Department of Dermatology, Quedlinburg

IPD SHARING:
Plan to Share IPD: No
patients/samples will be pseudonymized/anonymized